CLINICAL TRIAL: NCT01203033
Title: Prospective Pilot Study of Bone Marrow and Peripheral Blood Samples From Acute Myeloid Leukemia (AML) Patients to Characterize the Biologic Heterogeneity of the Disease Using Single Cell Network Profiling (SCNP)
Brief Title: Prospective Pilot Study of Bone Marrow and Peripheral Blood Samples From AML Patients to Characterize the Biologic Heterogeneity of the Disease Using Single Cell Network Profiling (SCNP)
Status: Completed | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Other Study IDs: WVU 1910
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; single cell network profiling; AML; SCNP
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AML patients: newly diagnosed or relapsed AML patients

SUMMARY:
Treatment options and clinical outcomes for acute myeloid leukemia (AML) have not improved for more than 40 years. AML patients are still suffering from receiving costly, ineffective chemotherapy treatments with very high chances of bad side effects. The purpose of this study is to take a look at leukemia cells to see if the investigators can learn what makes them up and makes them aggressive and hard to treat. We want to use this information to create new treatments that the investigators hope are more effective and less harmful for AML patients.

Newly diagnosed, relapsed or refractory (post induction therapy) AML patients that are 18 years of age or older will have bone marrow and blood samples taken for their regular AML treatment. When these tests are done during their treatment the investigators will need to get some extra blood and bone marrow to do this research. The patients will not be asked to have an extra needle stick or bone marrow biopsy to get these samples. The patients will have the same number of blood and bone marrow tests whether they participate in this study or not. We will only need to get about two teaspoons of blood and two teaspoons of bone marrow each time the patient has these tests during their regular AML treatment. The research the investigators do with these sample will not decide or change the care the patients get for their AML.

DETAILED DESCRIPTION:
The proposed study will be an open-label prospective investigation using fresh bone marrow and paired peripheral blood samples obtained from patients with AML starting at the time of diagnosis and including samplings at times of response assessment (CR and NR) continuing through relapse for responders and for other subsequent treatments including salvage therapy after resistance/relapse. Approximately 100 AML patients are expected to be enrolled. There is no extra marrow and blood sampling taken from patients who enroll into this study because we only study their marrow and blood when they undergo such sampling for routine medical needs. The SCNP results will not be used to guide or adjust current, or future, treatment for patients enrolled in this study and they will not be contacted regarding the study results.

Fresh whole bone marrow (5-10ml) and paired peripheral blood (5-10ml) will be collected from AML patients at participating institutions when these patients need marrow/blood tests prior to initiation of therapy, post each induction, post consolidation, at relapse and/or refractory, which is according to their standard care. When marrow cannot be obtained it is acceptable to collect only peripheral blood from the patient. Patient's demographic information, diagnosis, treatment option, outcome will be de-identified by the study PI. Samples must be collected in a standard 10 ml green top heparinized vacutainer labeled with sample de-identified ID, time, and date of collection. Samples will then be shipped to Nodality Inc. via FedEx in ambient temperature shipping kits on the same day. Nodality Inc. personnel will process the sample for study within 36 hours from collection. Leukemic blast SCNP will be conducted under the supervision of the researchers at Nodality Inc. and at facilities owned by Nodality Inc. Samples will be fractionated into bone marrow mononuclear cells (BMMC) or peripheral blood mononuclear cells (PBMC) and then aliquoted. All but one of these fractionated aliquots will be cryopreserved. The fresh, fractionated aliquot will be incubated with cytokines (e.g. interleukins, Flt3L), growth factors (e.g. SCF, GM-CSF and G-CSF), chemotherapeutic agents (e.g. cytarabine, ara- C, etoposide), and other modulators. Cells will then be fixed, permeabilized, and stained with antibodies that recognize extracellular markers (i.e. surface phenotypic markers such as clusters of differentiation, drug transporters, and receptors) in conjunction with intracellular activation-state specific epitopes (readouts) of designated signaling molecules. Subsequently, cells will be processed by multiparametric flow cytometry for SCNP. Blast populations will be defined by using combination of surface markers (CD33, CD34, CD38, CD45, CD11b) and approximately 30 different signaling nodes (paired modulator/readout e.g. Flt3L → phospho-Erk), depending on sample cell number (ideally 5-6 million; minimum 3 million). Signaling readouts will be evaluated in the total blast population, as well as within individual subpopulations, defined by CD33, CD34, CD 38, CD45, CD11b, and Side Scatter (SSC). Signaling readouts will be analyzed for each signaling node (univariate analysis) as well as a combination of nodes when the data set allows for multivariate analyses. In the "bridging" assay, cell surface markers and signaling readouts will be compared between fresh and cryopreserved AML samples including BMMC and PBMC when available in addition to BM samples.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, relapsed, or refractory (post induction therapy) AML patients age > 18
* For relapsed AML patients, previous treatment regimens received do not limit their eligibility to this study
* Patients enrolled will have no limitation as to the type of treatment they receive for their disease.
* Patient is able to give consent

Exclusion Criteria:

* AML-M3 patients
* AML patients age < 18
* AML patients in clinical remission
* AML patients who will not be able to receive diagnostic blood and marrow work up for any reason
* Patients who received allogeneic stem cell transplantation or autologous stem cell transplantation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed or relapsed AML patients at the Mary Babb Randolph Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To characterize the biologic phenotypes of leukemic blast cells in bone marrow and peripheral blood samples collected from AML patients during the natural history of the disease. | 3 years
To "bridge" assay performance between fresh and cryopreserved bone marrow and peripheral blood samples from AML patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: William Tse, MD, Principal Investigator — WVUCI - Mary Babb Randolph Cancer Center
Locations (1):
- MBRCC, West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No